CLINICAL TRIAL: NCT05156099
Title: A Pilot Study to Evaluate Anaesthetists' Ultrasound Scanning & Interpretation Performance for Ultrasound-guided Regional Anaesthesia - With & Without the Assistance of an Artificial Intelligence Device ScanNav Anatomy Peripheral Nerve Block
Brief Title: Clinical Performance Study: Evaluate Scanning & Interpretation Performance With & Without ScanNav Anatomy PNB
Acronym: PNB
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2021_AG_06
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Ultrasound Imaging of Anatomical Structures
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ScanNav Anatomy PNB unaided: The participants will be asked to perform clinically relevant tasks on multiple healthy volunteers while under observation by a subject matter expert (expert observer) who will assess participant performance without the device.
  Interventions: Device: Ultrasound Scanning; Device: Ultrasound Scanning - 2 months later
- ScanNav Anatomy PNB-aided: The participants will be asked to perform clinically relevant tasks on multiple healthy volunteers while under observation by a subject matter expert (expert observer) who will assess participant performance with the device.
  Interventions: Device: Ultrasound Scanning; Device: Ultrasound Scanning - 2 months later

INTERVENTIONS:
Device: Ultrasound Scanning — The participants will be asked to perform clinically relevant tasks on multiple healthy volunteers while under observation by a subject matter expert (expert observer) who will assess participant performance.
Device: Ultrasound Scanning - 2 months later — The participants will be asked to perform clinically relevant tasks on multiple healthy volunteers while under observation by a subject matter expert (expert observer) who will assess participant performance.

SUMMARY:
This is a single-centre, randomised, interventional prospective cohort study to be undertaken at offices of Intelligent Ultrasound Limited in Cardiff, United Kingdom.

DETAILED DESCRIPTION:
Current National Institute for Health and Care Excellence (NICE) guidance (NICE, 2009) supports the use of ultrasound-guidance for regional anaesthesia (UGRA) procedures as a consensus of clinical opinion agrees that nerve blocks are more successful and safer with ultrasound (US) guidance. Despite this, UGRA remains a difficult technique to master. This study will be used to determine whether ScanNav Anatomy PNB can support the performance of non-expert anaesthetist in UGRA scanning by highlighting key anatomical structures on the US image in real time.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study
3. Available to travel and attend the study day in person in Cardiff, UK
4. Medical professional (currently practicing anaesthetist or similar clinician) who is qualified to perform UGRA
5. Do not self-identify as an expert in the field of UGRA:

   1. Has not completed advanced training or hold a qualification (e.g., EDRA, MSc, MD, PhD) related to UGRA
   2. Does not regularly deliver anaesthesia for 'awake' surgery (excluding central neuraxial techniques)
   3. Does not teach on formal RA courses

Exclusion Criteria:

1. Aged <18 years of age
2. Unwilling or unable to provide informed consent
3. Expert in UGRA (see definition above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 24 participants will be recruited to represent the intended user population (anaesthetists qualified to perform UGRA, but non-experts in the field of regional anaesthesia), with an approximate 50/50 split between consultants and trainees.
  Potential study participants will be identified by approaching professional anaesthesia/anaesthetics societies, networks (e.g., Wales Regional Anaesthesia Group - South). Study participants will be required to attend one of the study assessment days at Intelligent Ultrasound head office in Cardiff, UK.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Correct identification of appropriate block site (at initial assessment and 2 months later) | 12 months
  Quantify the performance change associated with ScanNav Anatomy PNB during UGRA scanning: (for block regions of the upper limb, trunk, and lower limb).
  Correct identification of appropriate block site by participant [expert observer's opinion; Y/N]

SECONDARY OUTCOMES:
Time required to scan (at initial assessment and 2 months later) | 12 months
  Quantify the performance change associated with ScanNav Anatomy PNB during UGRA scanning: (for block regions of the upper limb, trunk, and lower limb) Time in seconds required for participant to scan [to obtain a satisfactory view of an appropriate block site, in the participant's opinion]
confidence in identifying an appropriate block site (at initial assessment and 2 months later) | 12 months
  Quantify the performance change associated with ScanNav Anatomy PNB during UGRA scanning: (for block regions of the upper limb, trunk, and lower limb)
  Participant confidence in identifying an appropriate block site [0 (no confidence] - 10 (total confidence)]
Correct identification of key structures (at initial assessment and 2 months later) | 12 months
  Quantify the performance change associated with ScanNav Anatomy PNB during UGRA scanning: (for block regions of the upper limb, trunk, and lower limb) Correct identification of key structures (including safety critical) at that block site by participant [expert observer's opinion; Y/N]
Expert observer's assessment (at initial assessment and 2 months later) | 12 months
  Quantify the performance change associated with ScanNav Anatomy PNB during UGRA scanning (for block regions of the upper limb, trunk, and lower limb) Expert observer's assessment of the participant's total scanning performance [0 (poor) - 10 (excellent)]
Quantify the change in incorrect identification of safety critical anatomical structures (at initial assessment and 2 months later) | 12 months
  Quantify the change in incorrect identification of safety critical anatomical structures associated with ScanNav Anatomy PNB during UGRA scanning (for block regions of the upper limb, trunk and lower limb), False positive/negative identification rates for blood vessels, nerves, pleura and peritoneum by participant [expert observer's opinion of participant judgement; Y/N]

CONTACTS AND LOCATIONS:
Overall Officials: James Bowness, Dr, Principal Investigator — OxSTaR, University of Oxford
Locations (1):
- Intelligent Ultrasound Limited, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowness JS, Macfarlane AJR, Burckett-St Laurent D, Harris C, Margetts S, Morecroft M, Phillips D, Rees T, Sleep N, Vasalauskaite A, West S, Noble JA, Higham H. Evaluation of the impact of assistive artificial intelligence on ultrasound scanning for regional anaesthesia. Br J Anaesth. 2023 Feb;130(2):226-233. doi: 10.1016/j.bja.2022.07.049. Epub 2022 Sep 8. PMID 36088136